CLINICAL TRIAL: NCT04507737
Title: Rapid Response Teams - How and Who? A Randomized Controlled Trial Examining the Composition of the RRT in a General Hospital
Brief Title: Rapid Response Teams - How and Who?
Acronym: RRT-Comp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pending
Record Dates: First submitted 2020-05-11; First posted 2020-08-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hospital Rapid Response Team; Early Warning Score; Intensive Care Units
MeSH Terms: interventions — Nurses

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Critical Care Outreach Team Model (Experimental): When a patient deteriorates and is in need of a Rapid Response Team, this arm will deploy a Critical Care Outreach Team Model consisting of an ICU-trained Nurse with the on-duty physician of the general ward and a nurse from the general ward.
  Interventions: Other: Rapid Response Team Composition_ ICU Nurse
- Medical Emergency team Model (No Intervention): When a patient deteriorates and is in need of a Rapid Response Team, this arm will deploy a Medical Emergency Team Model, consisting of an ICU-trained Doctor as well as an ICU-trained Nurse with the on-duty physician of the general ward and a nurse from the general ward.

INTERVENTIONS:
Other: Rapid Response Team Composition_ ICU Nurse — In case of deterioration a Rapid Response Team may be activated. We will be examining the composition of the teams alternating between a MET or a CCOT.
  Other Names: Rapid Response Team Composition - ICU Doctor + Nurse
  Arms: Critical Care Outreach Team Model

SUMMARY:
This will be an investigator initiated One-sided blinded Randomized Clinical Trial.

The study will examine the composition of the Rapid Response Team (RRT). the investigators will examine to see if a Critical Care Outreach Team (CCOT) consisting of an ICU-Nurse and a general ward physician and nurse are non-inferior to a Medical Emergency Team (MET) consisting of an ICU-Doctor and ICU Nurse as well as a general ward physician and nurse. The randomization will be done using an Analogue randomization sequence using sealed opaque envelopes with central randomization.The experimental intervention will be the CCOT. The statistical analyses will be done on the primary outcomes in the intention to treat population and on the secondary outcomes on an per-protocol basis exempting those with protocol violations.

DETAILED DESCRIPTION:
Trial design This trial is an investigator initiated, multi-centre, locally Randomized, one-side blinded trial of Nurse attended vs. Doctor attended RRT.

Randomization The patient will be screened for enrollment prior to the RRT leaving the ICU. A 1:1 randomization will occur at the time of call. The randomization will be with allocation concealment using a centrally randomized sequence at all participating sites. Due to time constraints the investigators will be using an analogue randomization sequence with sealed opaque envelopes. The Randomization sequence will be generated by a person independent of the project using Statistical software (SPSS or other like software) with a binary outcome of 0 or 1, where 0 will equal the control group and 1 will equal the intervention group. An independent group will then package sealed opaque envelopes in coherence with the sequence generated (controls will have blue cards, while interventions will be marked red). The sealed envelopes will be delivered to the primary investigator who will carry the responsibility of distributing these to the participating sites. When a patient is included the nurse will draw an envelope, open it, and sign the card which has been taken out. The local investigator or his/her delegate must on a daily basis collect and register the signed cards.

Blinding The allocation group is to be blinded for the investigators. As it is near impossible to blind the intervention for the clinicians the randomized allocation will not be blinded for the clinicians.

Members of the management committee (MC) will therefore not be involved in the daily clinical decision makings of the included patients. The outcome assessment will be blinded (i.e. registry-based assessment of interventions, evaluations, mortality, outcome and activation reasons). The statistical analyses will be with masked intervention groups i.e. coded as X/Y. And there will be done two conclusions, one defining x as the experimental group, and one assuming the opposite. The Steering Committee will be presented with two abstracts that must be accepted prior to breaking the bond.

If at anytime the investigators find it needed to investigate the results an Data Monitoring and Security Committee (DMSC) the members of the DMSC will remain blinded unless they 1) request unblinding or 2) find that an interim analysis provides strong indication of one intervention being beneficial or harmful.

Participant timeline The investigators will strive to enroll all patients fulfilling the inclusion criteria. Patients will receive either the experimental intervention of an ICU-Nurse attending the RRT, or the control of a Nurse and Doctor from the ICU attending the RRT. They will be followed up 30 days after RRT-event as well as 90- days post randomization. If another RRT-event occurs, within the same admission and within 30 days, another randomization will be performed, however the patient will only be included in the mortality comparison from the first randomization. If another RRT-event occurs within a new admission and within 30-days, the patient will receive another randomization however the patient will only be included in the mortality comparison from the first randomization. If another RRT-event occurs within a new admission after 30 days post randomization, the patient will receive a new randomization and will also be included in the mortality analysis twice.

Trial interventions Experimental intervention To ensure no dropout of data only MET-events where a MET-record is entered in the Electronic Medical Record (EMR) will be included.

The experimental intervention will be a MET-event attended only by an Intensive Care Unit Nurse, the team being led by the ward physician who is also responsible for treatment, even if this doctor is a junior doctor. All departments will be required to have a ward-physician attending a T-event in the trial period.

The ICU-nurse will be required to fill out an entry regarding the MET-event in the patients EMR, where details regarding the call may be registered Control intervention The control intervention will be standardized MET with both ICU doctor and ICU Nurse attending the patient. The ICU doctor will be team leader and the ward physician will be responsible for treatment as always.

The ICU doctor will be required to fill out an entry regarding the MET-event in the patients EMR, where details regarding the call may be registered Data collection Method Data will be obtained from the participants hospital files and national/regional/hospital registers (source data as defined per site, region and country) and by participant survey / interview and entered in the web-based REDCap database by trial investigators or their delegates. For participants transferred from a trial site to a non-trial site, data related to the outcomes will be collected according to national practice i.e. investigator contact to the relevant site or health-care registers.

Baseline variables are:

* Age
* Sex
* Time and Date of admission to hospital
* If applicable Time and Date of admission to ICU
* Time and Date of discharge
* Ward of RRT event
* Specialty responsible for the patient
* Admission cause

ELIGIBILITY:
Inclusion Criteria:

* Admitted to any general ward of the hospital AND
* Aged ≥ 18 years AND
* In need of RRT attention

Exclusion Criteria:

* Age < 18
* Admitted to the delivery ward
* Admitted to any ward in the anesthetic department

  * ICU
  * High Dependency Unit
  * Post Operation Department
  * Operating Theatre
  * Same Day Admissions - Surgery Ward
* Not admitted at the time of call

  * Evaluation track in Emergency department (prior to being seen by a doctor)
  * Out-Patient departments
  * X-ray department
* Any patient who cannot be randomized at the time of call

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
30-Day Mortality | up to 30 days
  Binary outcome measured via the patient Electronic Medical Records
In-Hospital Cardiac Arrest (IHCA) | up to 30 days
  Binary outcome measured via the patient Electronic Medical Records: defined as any IHCA post randomization and until discharge or 30 days post randomization
Unplanned Admission to the Intensive Care Unit | up to 30 days
  Binary outcome measured via the patient Electronic Medical Records. Defined as Admission to the ICU more than 24h Post randomization until discharge or 30 day post randomization
Unexpected Death | up to 30 days
  Binary outcome measured via the Patient Electronic Medical Records and National Register of deaths in the population. Defined as Any deaths post randomization until discharge or 30 days post randomization without treatment limitation being implemented during or 24 hours after the RRT, and without a "do not attempt resuscitation" order

SECONDARY OUTCOMES:
Activation of escape protocol | Through intervention completion, an average of 45 minutes
  Besides a few defined criteria the nurse may at any time activate the escape protocol and summon the ICU doctor to the patient immediately. If this is done at any time, it will be logged in the Electronic Medical Records and subsequently registered in the eCRF
90-day mortality | 90 days
  Binary outcome measured via the Patient electronic medical records.
Time Spent Bedside | Through intervention completion, an average of 45 minutes
  Continuous outcome measured via the Patient Electronic medical records - the MET-note. Defined in Minutes
Initiation of End of Life Care (EOL) | Maximum 30 days post randomization
  Binary outcome measured via the Patient Electronic Medical Records, defined as any treatment limitations involving cessation of all treatment, prescription of a safety/comfort package, No increase in treatment level - no ICU involvement and no MET involvement.
Score To Door Time | Through intervention completion, an average of 4 hours
  Continuous outcome calculated via the Patient Electronic medical records the MET-note, defined as the time from activation of the RRT until arrival at the ICU.
Survival until discharge | From date of admission until the date discharged up to 1 year.
  Binary outcome measured via the patient Electronic Medical Records
Length of Stay | From date of admission until discharged up to 1 year
  Continuous outcome measured via the Patient Electronic Medical records defined in Days, measured from admission date till discharge or death date.

OTHER OUTCOMES:
Activation reason | Through intervention completion, an average of 45 minutes
  Exploratory outcome regarding the reason for activating the MET
Interventions done by the RRT | Through intervention completion, an average of 45 minutes
  Exploratory outcome regarding the interventions done by the RRT
Outcomes from the RRT -event | Through intervention completion, an average of 45 minutes
  Exploratory outcome regarding the outcomes when the RRT-event is ending.
Evaluations by the RRT | Through intervention completion, an average of 45 minutes
  Exploratory outcome regarding the evaluations done by the RRT

CONTACTS AND LOCATIONS:
Locations (1):
- Nordsjællands Hospital, Hillerød, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Pending
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 9 months after finalized randomisation for 5 years